CLINICAL TRIAL: NCT05115201
Title: Effect of Antibiotics as an Adjuvant to Scaling and Root Planing on Systemic Inflammation in Patients With Periodontitis - A Randomized Clinical Trial.
Brief Title: Effect of Antibiotics on Systemic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Manpreet Kaur perio 2021
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis
Keywords: Anti-bacterial agents; inflammation; periodontitis
MeSH Terms: conditions — Periodontitis; Inflammation | interventions — Tooth Exfoliation; Root Planing; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (TG) (Experimental): Patients will be given amoxicillin and metronidazole, 500mg and 400mg respectively (AMX+MTZ) to be taken thrice daily for 7 days, as an adjuvant to scaling and root planing.
  Interventions: Procedure: Scaling and root planing with antibiotics
- Control group (CG) (Active Comparator): Patients will be treated with scaling and root planing only
  Interventions: Procedure: Scaling and root planing only

INTERVENTIONS:
Procedure: Scaling and root planing with antibiotics — Patients will be given amoxicillin and metronidazole, 500mg and 400mg respectively (AMX+MTZ) to be taken thrice daily for 7 days, as an adjuvant to scaling and root planing.
  Arms: Test group (TG)
Procedure: Scaling and root planing only — Patients will be treated with scaling and root planing
  Arms: Control group (CG)

SUMMARY:
Evidence support that pathogenic bacteria are not only responsible for periodontal destruction but also contributes to systemic inflammatory burden either directly or indirectly through increase in pro-inflammatory cytokines. Scaling and root planing (SRP) with or without local antibiotics contributes to reduced systemic inflammation. However, studies also reported insignificant changes in systemic inflammation after SRP. It may be due to incomplete control of periodontal inflammation. Systemic antibiotics proves to beneficial in treatment of severe periodontitis. Systemic antibiotics along with SRP results in improvement of vascular health and systemic inflammation. However, till date no study has been done to evaluate the role of systemic antibiotics as an adjunct to SRP on systemic inflammatory markers. In this randomized control study impact of adjunctive use of systemic antibiotics along with SRP on systemic inflammation would be assessed in periodontitis patients.

DETAILED DESCRIPTION:
Periodontitis is characterized by microbially-associated, host-mediated inflammation that results in loss of periodontal attachment. Periodontal bacteria possess a plethora of virulence factors that induce cells to produce inflammatory mediators at the gingival level.

Periodontitis is associated with bacteraemia that arises from perturbation of ulcerated periodontal tissues by simple acts of tooth brushing, eating and also during periodontal interventions disseminating whole bacteria and their products and toxins such as LPS. Virulence factors and bacteria itself interact with the host immune system and initiate inflammatory responses.

Moreover, bacteria may persist at distal sites disseminating virulence factors that act as soluble antigens thereby provocation leucocytes, endothelial cells and hepatocytes to respond to bacteria/virulence factors with secretion of pro-inflammatory immune mediators [cytokines, chemokines, C-reactive protein (CRP)]. With continued exposure, soluble antigens react with circulating specific antibody to form immune complexes that further amplify inflammation at sites of deposition.

In industrialized countries, approximately 50% of the adult population suffers from moderate or severe periodontitis. Basic periodontal therapy usually comprises mechanical debridement of the teeth. It is the disruption of biofilm, followed by lifelong maintenance therapy.

Traditional periodontal therapy involves elimination of periodontopathogens by mechanical debridement, such as scaling and root planing (SRP) and surgical procedures in conjunction with proper plaque control.

Because of the infective nature of periodontitis, pharmacologic agents have been advocated as adjuncts in the non-surgical treatment of periodontal infection. The rationale for the adjunctive use of antibiotics is to exert an antimicrobial effect at sites inaccessible to mechanical therapy, and possibly to suppress periodontal pathogens. Moreover, absence of specific periodontal pathogens seems to have a negative predictive value for further attachment loss. Therefore, one objective of periodontal treatment might be to suppress or eliminate certain subgingival periodontal pathogens. Adjunctive antibiotics have been suggested to improve treatment outcomes in patients with severe chronic periodontitis and aggressive periodontitis.

Because of amoxicillin and metronidazole's proven ability to suppress periodontal pathogens, such as A. actinomycetemcomitans and black pigmented bacteria from periodontitis lesions and other oral sites, it is the first choice of many clinicians, especially for the treatment of advanced A. actinomycetemcomitans-associated periodontitis. These pathogenic bacteria are not only restricted to oral cavity, but are associated with disease implication in other parts of the body.

Evidence support that pathogenic bacteria are not only responsible for periodontal destruction but also contributes to systemic inflammatory burden either directly or indirectly through increase in pro-inflammatory cytokines. Scaling and root planing with or without local antibiotics contributes to reduced systemic inflammation. However, studies also reported insignificant changes in systemic inflammation after SRP. It may be due to incomplete control of periodontal inflammation. Systemic antibiotics proves to beneficial in treatment of severe periodontitis. Systemic antibiotics along with scaling and root planing results in improvement of vascular health and systemic inflammation. However, till date no study has been done to evaluate the role of systemic antibiotics as an adjunct to scaling and root planing on systemic inflammatory markers.

In this randomized controlled clinical trial, impact of adjunctive use of systemic antibiotics along with scaling and root planing on systemic inflammation would be assessed in periodontitis patients.

Material and methods:

The present randomized clinical trial will be conducted in Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences, Rohtak. The study protocol is according to the ethical standards of Helsinki Declaration 1975 as revised in 2013.

Study population:

Periodontally healthy individuals (PH) and stage III periodontitis patients of age 35-45 years will be recruited from outpatient department of Periodontics and Oral Implantology. The patients will be enrolled after obtaining an informed consent.

Experimental design: This randomized clinical trial consists of two parallel groups based intervention in periodontitis patients:

Periodontal parameters:

At baseline, periodontal parameters plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing pocket depth (PPD), clinical attachment loss (CAL) will be assessed at six sites (disto-buccal, mid-buccal, mesio-buccal, mesio-lingual, mid-lingual and disto-lingual) per tooth excluding third molars in all groups. Periodontal inflamed surface area (PISA) will then be calculated. Periodontal examination would again be done during recall visit after 2nd month in test group (TG) and control group (CG).

Periodontal therapy:

After recording periodontal parameters at baseline, oral hygiene instructions would be given and scaling and root planing (SRP) would be done in both treatment groups (TG and CG). TG will be given amoxicillin and metronidazole, 500mg and 400mg respectively (AMX+MTZ) to be taken thrice daily for 7 days. Patients will inform about any self-perceived side-effects of the medications. Any adverse effects from antibiotic intake and compliance, as reported by patients, will be recorded throughout the study period. TG and CG would be recalled after 1stand 2nd month of SRP. At recall visit after 1 month, oral hygiene instructions will be re-enforced and supportive periodontal therapy would be provided.

Blood collection and serum analysis:

For assessing markers of systemic inflammation, serum samples will be collected from venipuncture in antecubital fossa after an overnight fasting.

Serum samples would be analyzed for systemic markers at baseline and after 2 months of periodontal treatment in TG and CG.

Parameter of systemic inflammation that would be assessed:

• High sensitive C-reactive protein (hs CRP)

Blood parameters that would be assessed: Total leukocyte count(TLC), differential leukocyte count (DLC), neutrophil lymphocyte ratio, platelet count, mean platelet volume (MPV), platelet distribution width (PDW), platelet-to-lymphocyte ratio (PLR), red blood cell count (RBC), hemoglobin (Hb), hematocrit (Hct), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW)

Blood parameters that would be assessed: triglyceride (TG), total cholesterol (TC), low-density lipoprotein cholesterol (LDL), high-density lipoprotein cholesterol (HDL), very low-density lipoprotein cholesterol (VLDL)

Anthropometric parameter that would be measured: Body Mass Index (BMI) calculated as weight/height2 (Kg/m2) at baseline.

ELIGIBILITY:
Inclusion Criteria:

* • Systemically healthy individuals

  * Presence of at least 20 teeth excluding third molars.
  * PH individuals defined as <10% bleeding sites with probing depths ≤3mm.
  * Periodontitis criteria:

Stage III periodontitis with ≥30% teeth involved and bleeding on probing with >30% sites involved.

Exclusion Criteria:

* Confirmed or assumed allergies or hypersensitivity reactions to amoxicillin and/or metronidazole.
* Alcohol consumers.
* History of systemic medication affecting the periodontal conditions, e.g. steroids, immune suppressants, antibiotics, anti-inﬂammatory drugs, statins, lipid lowering drugs, anti-convulsants, anti-coagulants, anti-hypertensives or any other host modulatory drugs within 6 months of commencing the study.
* Had received any periodontal treatment in the previous 12 months.
* Undergoing or require an extensive dental or orthodontic treatment.
* Pregnant or breastfeeding women.
* Current or former users of tobacco in any form.

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
High senstivity C-reactive protein (hsCRP) | 2 months
  For assessing marker of systemic inflammation, serum samples will be collected from venipuncture in antecubital fossa after an overnight fasting.

CONTACTS AND LOCATIONS:
Overall Officials: MANPREET KAUR, MDS, Principal Investigator — Post Graduate Institute of Dental Sciences, Rohtak
Locations (1):
- Sanjay Tewari, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No